CLINICAL TRIAL: NCT06426836
Title: Pediatric Antibiotic Dosing in Extracorporal Membrane Oxygenation
Brief Title: Pediatric Antibiotic Dosing in Extracorporal Membrane Oxygenation (PADECMO)
Acronym: PADECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EC 2015/0529
Record Dates: First submitted 2022-05-13; First posted 2024-05-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetics; Amoxicillin-clavulanate; Piperacillin-tazobactam; Meropenem; Cefazolin; Teicoplanin; Vancomycin; Ciprofloxacin; Amikacin
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Blood Specimen Collection; Piperacillin, Tazobactam Drug Combination; Meropenem; Cefazolin; Vancomycin; Teicoplanin; Ciprofloxacin; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Amoxicillin-clavulanate (Other): Patients receiving amoxicillin-clavulanate as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Amoxicillin-clavulanate
- Piperacillin-tazobactam (Other): Patients receiving piperacillin-tazobactam as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Piperacillin-tazobactam
- Meropenem (Other): Patients receiving meropenem as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Meropenem
- Cefazolin (Other): Patients receiving cefazolin as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Cefazolin
- Vancomycin (Other): Patients receiving vancomycin as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Vancomycin
- Teicoplanin (Other): Patients receiving teicoplanin as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Teicoplanin
- Ciprofloxacin (Other): Patients receiving ciprofloxacin as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Ciprofloxacin
- Amikacin (Other): Patients receiving amikacin as part of routine clinical care. Study procedure: blood sampling
  Interventions: Other: Amikacin

INTERVENTIONS:
Other: Amoxicillin-clavulanate — blood sampling in patients receiving amoxicillin-clavulanate as part of routine clinical care
  Other Names: Blood sampling
  Arms: Amoxicillin-clavulanate
Other: Piperacillin-tazobactam — blood sampling in patients receiving piperacillin-tazobactam as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Piperacillin-tazobactam
Other: Meropenem — blood sampling in patients receiving meropenem as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Meropenem
Other: Cefazolin — blood sampling in patients receiving cefazolin as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Cefazolin
Other: Vancomycin — blood sampling in patients receiving vancomycin as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Vancomycin
Other: Teicoplanin — blood sampling in patients receiving teicoplanin as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Teicoplanin
Other: Ciprofloxacin — blood sampling and urine sampling in patients receiving ciprofloxacin as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Ciprofloxacin
Other: Amikacin — blood sampling in patients receiving amikacin as part of routine clinical care.
  Other Names: Blood sampling
  Arms: Amikacin

SUMMARY:
Pharmacokinetics of antibiotics in critically ill neonates, infants and children on extracorporeal membrane oxygenation (ECMO).

DETAILED DESCRIPTION:
The study will investigate whether - with the current dosing regimens of meropenem, piperacillin-tazobactam, amoxicillin-clavulanate, cephazolin, vancomycin, amikacin, teicoplanin and ciprofloxacin - pharmacodynamic targets are attained in a national multicentric clinical setting in pediatric patients on ECMO.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the pediatric intensive care unit or cardiac intensive care unit
* patient age : 1,8 kg-15 years
* patient receiving antibiotic treatment (piperacillin-tazobactam, meropenem, amoxicillin-clavulanate, cephazolin, vancomycin, teicoplanin, ciprofloxacin, amikacin)
* intra-arterial or intravenous access other than the drug infusion line available for blood sampling (arterial line is preferred)
* extracorporeal membrane oxygenation circuit

Exclusion Criteria:

* no catheter in place for blood sampling
* absence of parental/patient consent
* known hypersensitivity to beta-lactam antibiotics and ciprofloxacin

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2016-08-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Amoxicillin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens on extracorporeal membrane oxygenation in steady-state conditions
Cefazolin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens on extracorporeal membrane oxygenation in steady-state conditions
Meropenem: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens on extracorporeal membrane oxygenation in steady-state conditions
Piperacillin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens on extracorporeal membrane oxygenation in steady-state conditions
Amoxicillin, piperacillin, meropenem, cefazolin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens before or after extracorporeal membrane oxygenation in steady-state conditions
Cefazolin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens before or after extracorporeal membrane oxygenation in steady-state conditions
Meropenem: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens before or after extracorporeal membrane oxygenation in steady-state conditions
Piperacillin: probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) of the micro-organism | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens before or after extracorporeal membrane oxygenation in steady-state conditions
Ciprofloxacin: probability of target attainment with the target being the free Area-under the Concentration-Time Curve over Minimal Inhibitory Concentration ratio (fAUC/MIC) | up to 1 month
  % of patients for whom a fAUC/MIC target>86 is achieved with the current dosing regimen off extracorporeal membrane oxygenation in steady-state conditions
Vancomycin: probability of target attainment with the target being the Area-under the Concentration-Time Curve over Minimal Inhibitory Concentration (AUC/MIC) | up to 1 month
  % of patients in whom a AUC/MIC target 400-600 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in steady-state conditions
Teicoplanin: probability of target attainment with the target being a mimimal trough concentration | up to 1 month
  % of patients in whom a trough concentration between 20 to 30 mg/L is achieved with the current dosing regimen on extracorporeal membrane oxygenation in steady-state conditions
for teicoplanin: probability of target attainment with the target being an Area-under the Concentration-Time Curve over Minimal Inhibitory Concentration Ratio (AUC/MIC) | up to 1 month
  % of patients in whom an AUC/MIC of 900 is achieved with the current dosing regimen before or after extracorporeal membrane oxygenation in steady-state conditions
for amikacin: probability of target attainment with the target being a peak concentration over Minimal Inhibitory Concentration ratio (peak/MIC) | up to 1 month
  % of patients in whom a target peak/MIC ratio of 8 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in steady-state conditions
Amikacin: probability of toxicity threshold attainment with a target being a minimal trough concentration | up to 1 month
  % of patients in whom the threshold for toxicity concentration>5 mg/L is achieved with the current dosing regimen on extracorporeal membrane oxygenation in steady-state conditions
Amikacin: probability of toxicity threshold attainment with a target being a minimal trough concentration | up to 1 month
  % of patients in whom the threshold for toxicity concentration>5 mg/L is achieved with the current dosing regimen before or after extracorporeal membrane oxygenation in steady-state conditions
Amikacin: probability of target attainment with the target being a free Area-under-the-Concentration-Time Curve over Minimal Inhibitory Concentration ratio (AUC/MIC) | July 2026
  % of patients in whom a target fAUC/MIC ratio of 399 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in steady-state conditions
Amikacin: probability of target attainment with the target being a free Area-under-the-Concentration-Time Curve over Minimal Inhibitory Concentration ratio (AUC/MIC) | July 2026
  % of patients in whom a target fAUC/MIC ratio of 399 is achieved with the current dosing regimen before or after extracorporeal membrane oxygenation in steady-state conditions

SECONDARY OUTCOMES:
Risk factors for underdosing during extracorporeal membrane oxygenation for beta-lactam antibiotics | up to 1 month
  The impact of demographic, clinical characteristics and ECMO equipment characteristics on the risk of underdosing and overdosing will be investigated. The pharmacokinetic/pharmacodynamic target that is used is a percentage of time during which the unbound concentration remains above the Minimal Inhibitory Concentration (MIC) of the micro-organism of at least 50% and a maximum concentration of 10 x MIC
Risk factors for underdosing during extracorporeal membrane oxygenation for ciprofloxacin | up to 1 month
  The impact of demographic, clinical characteristics and ECMO equipment characteristics on the risk of underdosing and overdosing of ciprofloxacin will be investigated. The pharmacokinetic/pharmacodynamic target that is used is a free Area-under the concentration-Time Curve of 86
Risk factors for under-and overdosing during extracorporeal membrane oxygenation for vancomycin | up to 1 month
  The impact of demographic, clinical characteristics and ECMO equipment characteristics on the risk of underdosing and overdosing of vancomycin will be investigated. The pharmacokinetic/pharmacodynamic target that is used is a free Area-under the concentration-Time Curve of 200 to 300
Risk factors for underdosing during extracorporeal membrane oxygenation for teicoplanin | up to 1 month
  The impact of demographic, clinical characteristics and ECMO equipment characteristics on the risk of underdosing and overdosing of teicoplanin will be investigated. The pharmacokinetic/pharmacodynamic target that is used is an Area-under the concentration-Time Curve of 900
Risk factors for under-and overdosing during extracorporeal membrane oxygenation for amikacin | up to 1 month
  The impact of demographic, clinical characteristics and ECMO equipment characteristics on the risk of underdosing and overdosing of amikacin will be investigated. The pharmacokinetic/pharmacodynamic target that is used is a peak over Minimal Inhibitory Concentration Ratio of 8 to 10, trough concentration below 5 mg/L and Area under the Concentration Time Curve/MIC>399
Beta-lactam antibiotics (amoxicillin, piperacillin, meropenem, cefazolin): probability of target attainment with target the % of time during which the unbound drug concentration remains above the Minimal Inhibitory Concentration (fT>MIC) | up to 1 month
  % of patients for whom a target of fT>MIC of 50% is achieved with current dosing regimens on extracorporeal membrane oxygenation in first dose conditions
Ciprofloxacin: probability of target attainment with the target being the free Area-under the Concentration-Time Curve over Minimal Inhibitory Concentration ratio (fAUC/MIC) | up to 1 month
  % of patients for whom a fAUC/MIC target>86 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in first-dose conditions
Vancomycin: probability of target attainment with the target being the Area-under the Concentration-Time Curve over Minimal Inhibitory Concentration (AUC/MIC) | up to 1 month
  % of patients in whom a AUC/MIC target 400-600 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in first-dose conditions
Teicoplanin: probability of target attainment with the target being a mimimal trough concentration | up to 1 month
  % of patients in whom a trough concentration between 20 to 30 mg/L is achieved with the current dosing regimen on extracorporeal membrane oxygenation in first-dose conditions
Amikacin: probability of target attainment with the target being a peak concentration over Minimal Inhibitory Concentration ratio (peak/MIC) | up to 1 month
  % of patients in whom a target peak/MIC ratio of 8 is achieved with the current dosing regimen on extracorporeal membrane oxygenation in first-dose conditions
Amikacin: probability of toxicity threshold attainment with a target being a minimal trough concentration | up to 1 month
  % of patients in whom the threshold for toxicity concentration>5 mg/L is achieved with the current dosing regimen on extracorporeal membrane oxygenation in first-dose conditions

CONTACTS AND LOCATIONS:
Overall Officials: Annick de Jaeger, MD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - Queen Fabiola Children's University Hospital, Brussels, Brussels Capital
  - University Hospital, Ghent
  - Universitair hospital, Leuven

IPD SHARING:
Plan to Share IPD: Undecided